CLINICAL TRIAL: NCT03180892
Title: Non-immune Related Hypothyroidism in Iodine Sufficient Area
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hoon Chung, M.D., Ph.D., Samsung Medical Center
Other Study IDs: 2017-05-149
Record Dates: First submitted 2017-06-02; First posted 2017-06-08 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Hypothyroidism
Keywords: Iodine; thyroid peroxidase antibody
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The investigators did not apply any intervention for the participants. — The investigators did not apply any intervention for the participants.

SUMMARY:
Background: Autoimmune hypothyroidism has been regarded as the most common cause of primary hypothyroidism in iodine sufficient area and has relationship with excess iodine induced hypothyroidism. However, non-immune related hypothyroidism and its relationship with excess iodine have been rarely evaluated.

Objective: Therefore, the investigators planned to calculate proportion of non-immune related hypothyroidism and relationship with iodine intake using nationwide data from Korea National Health and Nutrition Examination Survey (KNHANES) 2013-2015.

Design:

1. Korea National Health and Nutrition Examination Survey VI (2013 to 2015) - The national data - which is the government designated statistics (Approval No. 117002 ) of South Korea based on the Article 17 of the National Health Promotion Act - were used. The survey was approved by the Institutional Review Board of the Korea Centers for Disease Control and Prevention, and provides only non-identified measures for academic research purposes.
2. The participants who were examined for thyroid stimulating hormone, free thyroxine, thyroid peroxidase antibody (TPO Ab), and urine iodine concentration (UIC) were included.
3. The proportion of immune related and non-immune related hypothyroidism was evaluated. Demographic variables and severity of hypothyroidism were compared between the two groups. To analyze iodine effect on hypothyroidism in TPO Ab positive or negative population, prevalence of hypothyroidism were assessed in each TPO Ab negative and positive population according to UIC subgroups.
4. This study protocol was approved by IRB of SMC (2017-05-149).

ELIGIBILITY:
Inclusion Criteria:

* examined for thyroid stimulating hormone, free thyroxine, thyroid peroxidase antibody (TPO Ab), and urine iodine concentration (UIC)

Exclusion Criteria:

* already have a thyroid disease(benign thyroid diseases or thyroid cancer).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators used a dataset from the KNHANES VI (2013 to 2015), a nationwide, cross-sectional survey of the Korean population for surveillance of health and nutritional status. The survey used stratified, multistage clustered probability sampling to select a representative sample of the civilian non-institutionalized Korean population. Research subjects were selected through two-stage stratified cluster sampling using population and housing census data. The investigators included the subjects who were examined for TSH, FT4, TPO Ab, and UIC. Subjects previously diagnosed with benign thyroid diseases or thyroid cancer were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 6564 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The weighted proportion of non-immune related hypothyroidism | 3 years
  Hypothyroidism with TPO Ab negative

IPD SHARING:
Plan to Share IPD: Yes
This data is national data of Korea. It is already possible to use the data freely only for the purpose of academic research and the like.